CLINICAL TRIAL: NCT05268549
Title: Independent Risk Factors Analysis and Model Construction For Recurrence After Radiofrequency/Microwave Ablation of Colorectal Cancer With Liver Metastases: a Retrospective, Multicenter Trial
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The Central Hospital of Lishui City (Other)
Collaborators: Zhejiang Cancer Hospital (Other); Zhejiang University (Other); First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: ZJLS-KLDMIR-22005
Record Dates: First submitted 2022-02-10; First posted 2022-03-07 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-03

CONDITIONS: Colorectal Cancer With Liver Metastases
Keywords: colorectal cancer with liver metastases; Radiofrequency/Microwave; Recurrence
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a retrospective, multicenter clinical study. The main objective is to analyze the risk factors affecting the recurrence of colorectal cancer patients with liver metastases who received radiofrequency/microwave ablation. Finally, we will construct a recurrence risk prediction model based on the risk factors and validated the model.

ELIGIBILITY:
Inclusion Criteria:

1. Age：older than 18 years；
2. Patients with a single tumor diameter ≤5cm, no more than 3 tumor nodules, and the largest tumor diameter ≤3cm；
3. Absence of vessel, bile duct and adjacent organ invasion and distant metastasis;
4. The primary tumor of colorectal cancer has been resected, the liver metastases cannot be resected or the patient is unwilling to undergo surgery (clinical or pathological confirmation);
5. Normal coagulation status and liver function child-pugh A or B;
6. Liver metastases have not received other antitumor therapy after radiofrequency/microwave therapy (before disease progression);
7. Routine laboratory tests were performed before the first RF/microwave treatment;
8. Follow up for more than 12 months;
9. Obtained free informed consent.

Exclusion Criteria:

1. Large tumor, or diffuse intrahepatic metastasis;
2. Accompanied by vascular tumor thrombus or invasion of adjacent organs;
3. The primary tumor of colorectal cancer has not been resected, with extrahepatic metastasis;
4. Uncorrectable coagulation dysfunction and severe blood abnormalities, those with severe bleeding tendency;
5. Intractable massive ascites, cachexia;
6. Active infection, especially inflammation of the biliary system;
7. Severe liver, kidney, heart, lung, brain and other major organ failure;
8. Patients with impaired consciousness or unable to cooperate with treatment;
9. Missing follow-up data.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This is a multicenter study. Patients from Lishui Central Hospital of Zhejiang Province, Zhejiang Cancer Hospital, the First Affiliated Hospital of Zhejiang University, the Second Affiliated Hospital of Zhejiang University, and the First Affiliated Hospital of Wenzhou Medical University who meet the above criteria will be included in this study
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-03-12 (Estimated); Primary Completion 2022-05-12 (Estimated); Study Completion 2022-08-12 (Estimated)

PRIMARY OUTCOMES:
The first recurrence of colorectal cancer with liver metastasis (CRLM) after radiofrequency/microwave ablation, assessed up to 18 months | Time from enrollment to disease recurrence, assessed up to 18 months
  The first recurrence of colorectal cancer with liver metastasis (CRLM) after radiofrequency/microwave ablation, assessed up to 18 months

SECONDARY OUTCOMES:
Patients with colorectal cancer with liver metastases (CRLM) developed new metastases after radiofrequency/microwave ablation,assessed up to 18 months | Time from enrollment to developed new metastases, assessed up to 18 months
  Patients with colorectal cancer with liver metastases (CRLM) developed new metastases after radiofrequency/microwave ablation,assessed up to 18 months

IPD SHARING:
Plan to Share IPD: Yes
Statistical analysis plan, informed consent form, and clinical study report can be shared with other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within six months after the trial is completed.
Access Criteria: Shared data is not available for downloading, but can only be browsed. To download the data, you must contact the researchers. Shared data does not provide any private information of the participants.